CLINICAL TRIAL: NCT03455478
Title: Shanghai Eye Study for Adults
Acronym: SESA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: YFZX2018001
Record Dates: First submitted 2018-02-10; First posted 2018-03-06 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Blindness,Visual Impairment, Refractive Error, Cataract, High Myopia, Aging
MeSH Terms: conditions — Blindness; Vision Disorders; Refractive Errors; Cataract | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- corrected refractive error (Experimental)
  Interventions: Device: spectacles
- uncorrected refractive error (No Intervention)

INTERVENTIONS:
Device: spectacles — dispending spectacles for uncorrected refractive error
  Arms: corrected refractive error

SUMMARY:
Blindness and visual impairment severely impact the visual health and life quality of people, particularly the 2.566 million senior citizens aged at 65 and above in Shanghai. The main reason is uncorrected refractive error, of which, 62.1% can be solved through refractive correction. For this reason, the uncorrected refractive errors of 154,000 senior citizens in Shanghai can be taken as a priority among the public health issues to prevent blindness. Now, with the aim to reduce the prevalence rate of blindness and visual impairment, it is planned to establish a public health service mechanism in terms of refractive error screening and correction for the elderly by relying on Shanghai's three-level (city-district-community) eye diseases prevention network, using proper refractive correction technology, and moving related services forward to communities in order to screen, identity, and correct blindness and visual impairment caused by refractive errors as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* shanghai residents aged ≥18 years old

Exclusion Criteria:

* cognitive and/or mobility disorders; non-shanghai residents; younger than 18 years old.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
best-corrected visual acuity (BCVA) | 5 years
  the prevalence of blindness and visual impairment
cataract surgery rate | 5 years
  cataract surgery rate of Shanghai older people
cataract surgery coverage rate | 5 years
  cataract surgery coverage rate of Shanghai cataract patients
visual impairment caused by high myopia | 5 years
  observing the rate of visual impairment caused by high myopia

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided